CLINICAL TRIAL: NCT04625439
Title: Personality and Cancer Care Study: Examining the Effects of a Personality Feedback Intervention in Adults With Cancer
Brief Title: Personality and Cancer Care Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Responsible Party: Principal Investigator, Laura Perry, Principal Investigator, Tulane University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020-909
Record Dates: First submitted 2020-11-03; First posted 2020-11-12 (Actual); Last update posted 2021-03-02 (Actual); Status verified 2021-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personality Feedback (Experimental): The intervention arm will read about the Five-Factor model and receive a feedback report with individualized personality results and self-management recommendations.
  Interventions: Behavioral: Personality Feedback Self-Management Intervention
- No-feedback Control (No Intervention): The control arm will read about the Five-Factor model but will not receive feedback or their personality results until after the study.

INTERVENTIONS:
Behavioral: Personality Feedback Self-Management Intervention — The intervention is a personality feedback report that will tell participants whether they scored low (bottom third), average (middle third), or high (top third) on each of the five factor personality characteristics based on gender-matched norms. In addition to a description of general tendencies based on their level of each personality trait, the feedback will include information about how scoring in a given category may relate to an individual's cancer self-management or healthcare decision making. The feedback for each personality trait will include recommendations for how to improve key outcomes.
  Arms: Personality Feedback

SUMMARY:
This randomized clinical trial will test whether giving an individualized personality feedback report to adults with a history of cancer can improve their self-awareness, confidence in managing their illness, and mood.

DETAILED DESCRIPTION:
This will be a randomized clinical trial examining whether a personality feedback intervention can improve three outcomes in an online sample of adults with cancer: 1) self-awareness, 2) self-efficacy for managing aspects of their illness, and 3) mood. The study will occur in a single 30-minute online session conducted in Qualtrics, with a pre-post randomized design. Participants will respond to a baseline survey including a measurement of the Five-Factor Personality Model and measures of the 3 outcomes of interest, followed by random assignment to either an intervention group or control group. Both groups will read a brief description of the Five-Factor Model of Personality. Those randomized to the intervention group will also receive an individualized feedback report containing their personality results on each of the five personality factors and recommendations for cancer self-management based on these results. After reading the personality information, participants will respond to the outcome measures again in a post-intervention survey. Control participants will receive their individualized personality feedback reports after the study is complete.

ELIGIBILITY:
Inclusion Criteria:

* consent to participate
* at least 18 years old (self-reported)
* have a current or past cancer diagnosis (self-reported)

Exclusion Criteria:

* under 18 years old (self-reported)
* indicate that they have no known history of cancer (self-reported)
* unable to read or understand English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 419 (Actual)
Dates: Start 2020-11-18 (Actual); Primary Completion 2021-02-08 (Actual); Study Completion 2021-02-08 (Actual)

PRIMARY OUTCOMES:
Self-Awareness Outcomes Questionnaire - Change Score | pre-intervention and immediately post-intervention.
  Participants' current state-level self-awareness will be assessed with a modified 6-item short form of the Reflective Self-Development subscale included in the Self-Awareness Outcomes Questionnaire (SAOQ). Participants rate each item from 1 to 5, and a total score will be calculated by summing participants responses to each item. The total score at each time point will range from 6 to 30, with higher scores indicating higher levels of self-awareness. The difference score from pre-intervention to post-intervention will be used in analyses, with higher scores indicating a greater increase in self-awareness.

SECONDARY OUTCOMES:
PROMIS Self-Efficacy for Managing Chronic Conditions - Change Score | pre-intervention and immediately post-intervention.
  Participants will respond to three 4-item custom short forms from the Patient-Reported Outcomes Measurement Information System (PROMIS) Self-efficacy for Managing Chronic Conditions Domain: 1) self-efficacy for managing emotions, 2) self-efficacy for managing symptoms, and 3) self-efficacy for managing medications and treatment. Each item is rated from 1 to 5, with raw scores on a summated total scale for each subscale ranging from 4 to 20. Each subscale's raw total score will be converted to a T-score, and a mean composite T-score across the 3 subscales will be calculated for each time point. Higher scores indicate higher levels of self-efficacy for managing their illness. For analyses, the difference in the mean T-score from pre-intervention to post-intervention will be computed, with higher scores indicating a greater increase in self-efficacy for managing their illness.
PANAS Positive Affect Subscale - Change Score | pre-intervention and immediately post-intervention.
  The 10-item positive affect scale from the Positive and Negative Affect Schedule (PANAS) will be used to assess current mood. Participants rate each item from 1 to 5, and a total summated scale score will range from 10 to 50, with higher scores indicating higher levels of positive affect. For analyses, the difference score from pre-intervention to post-intervention will be calculated, with higher scores indicating a greater increase in positive mood.

CONTACTS AND LOCATIONS:
Overall Officials: Laura M Perry, MS, Principal Investigator — Tulane University
Locations (1):
- Tulane University, New Orleans, Louisiana, United States

REFERENCES:
- [Derived] Perry LM, Mossman B, Garcia SF, Kircher SM, Dunn A, Alonzi S, Easwar S, Hoerger M. Personality Feedback With Tailored Self-Care Recommendations Improves Self-Efficacy for Cancer Management: A Randomized Controlled Trial. Psychooncology. 2024 Nov;33(11):e70023. doi: 10.1002/pon.70023. PMID 39547948